CLINICAL TRIAL: NCT01998152
Title: The Effect of Individualized NUTritional Counselling on Muscle Mass and Treatment Outcome in Patients With Metastatic COLOrectal Cancer Undergoing Chemotherapy: the COLONUT Study
Brief Title: Individualized Nutritional Counselling During Chemotherapy for Colorectal Cancer (COLONUT)
Acronym: COLONUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, M.A.E van Bokhorst - de van der Schueren, Dr., Senior Investigator dietetics and nutrition sciences Vumc, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013230
Record Dates: First submitted 2013-11-11; First posted 2013-11-28 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Stage IV Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nutritional counseling (Experimental): Individualized nutritional counselling by a registered dietitian
  Interventions: Procedure: Nutritional counseling
- No intervention (No Intervention): Usual nutritional care by the oncologist. A dietitian is only involved when serious nutritional problems occur.

INTERVENTIONS:
Procedure: Nutritional counseling — Patients in the intervention-arm will receive individualized nutritional counseling by a registered dietitian during standard treatment with chemotherapy. The main goals of the nutritional intervention will be to enable every patient to achieve sufficient protein and energy intake with attention for sufficient intake of micronutrients and a sufficient physical activity level.
  Arms: Nutritional counseling

SUMMARY:
The purpose is to study the effect of individualized nutritional counselling compared to usual nutritional care on cross-sectional muscle area in patients with stage IV colorectal cancer during first line chemotherapy. Secondary, effect on total lean body mass, treatment intensity, physical functioning, quality of life and survival will be studied.We hypothesize that patients in the intervention arm benefit from individualized nutritional counseling.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Stage IV colorectal cancer
* Scheduled for treatment with first line chemotherapy, either CAPOX(-B), FOLFOX(-B) or capecitabine(-B)
* CT scan suitable for evaluating muscle mass at L3 level
* Understanding of the Dutch language
* Able and willing to give written informed consent

Exclusion Criteria:

* Chemotherapy in the previous three months
* WHO performance status ≥ 3
* Long-term high dose of corticosteroids: ≥ three weeks ≥ ten milligram prednisolon or equivalent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2013-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Change in skeletal muscle area (cm2) between individualized nutritional counselling versus usual nutritional care | During 9 weeks of first line chemotherapy
  will be measured with SliceOmatic software V5.0 (Tomovision) with use of routinely conducted CT scans for diagnostic and disease evaluation purposes

SECONDARY OUTCOMES:
Change in total body lean body mass and segmental lean body mass (DEXA) in patients with stage IV colorectal cancer during 9 weeks of first line chemotherapy between individualized nutritional counseling versus usual nutritional care | During 9 weeks of first line chemotherapy
Change in skeletal muscle area in patients with stage IV colorectal cancer during 20 weeks of first line chemotherapy between individualized nutritional counseling.versus usual nutritional care. | During 20 weeks of first line chemotherapy
  Change in skeletal muscle area (cm2) between individualized nutritional counselling versus usual nutritional care
Composite of treatment toxicity, treatment intensity, treatment outcome, survival, physical functioning, quality of life and hand grip strength of both study arms | During 9 weeks and during 20 weeks of first line chemotherapy
Associations of (changes in) muscle area with (changes in) mid-upper arm muscle circumference, whole body fat free mass (BIA) and whole body lean body mass (DEXA). | During 9 weeks of first line chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: M.A.E de van der Schueren, Dr., Principal Investigator — Amsterdam UMC, location VUmc
Locations (5):
- Netherlands (5):
  - VU Medical Center, Amsterdam
  - Amphia Hospital, Breda
  - Reinier de Graaf, Delft
  - Ziekenhuis Gelderse Vallei, Ede
  - Spaarne hospital, Hoofddorp

REFERENCES:
- [Derived] van der Werf A, Langius JAE, Beeker A, Ten Tije AJ, Vulink AJ, Haringhuizen A, Berkhof J, van der Vliet HJ, Verheul HMW, de van der Schueren MAE. The effect of nutritional counseling on muscle mass and treatment outcome in patients with metastatic colorectal cancer undergoing chemotherapy: A randomized controlled trial. Clin Nutr. 2020 Oct;39(10):3005-3013. doi: 10.1016/j.clnu.2020.01.009. Epub 2020 Jan 29. PMID 32037284
- [Derived] van der Werf A, Blauwhoff-Buskermolen S, Langius JA, Berkhof J, Verheul HM, de van der Schueren MA. The effect of individualized nutritional counseling on muscle mass and treatment outcome in patients with metastatic colorectal cancer undergoing chemotherapy: a randomized controlled trial protocol. BMC Cancer. 2015 Mar 5;15:98. doi: 10.1186/s12885-015-1092-5. PMID 25884881